CLINICAL TRIAL: NCT00118352
Title: Campath (Alemtuzumab) Dose Escalation, Low-Dose TBI and Fludarabine Followed by HLA Class II Mismatched Donor Stem Cell Transplantation for Patients With Hematologic Malignancies: A Multicenter Trial
Brief Title: Alemtuzumab, Fludarabine Phosphate, and Total-Body Irradiation Followed by Cyclosporine and Mycophenolate Mofetil in Treating Patients Who Are Undergoing Donor Stem Cell Transplant for Hematologic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Brenda Sandmaier, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1959.00; NCI-2009-01496 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1959.00 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); P01CA018029 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Atypical Chronic Myeloid Leukemia, BCR-ABL1 Negative; Childhood Acute Lymphoblastic Leukemia in Remission; Childhood Acute Myeloid Leukemia in Remission; Childhood Burkitt Lymphoma; Childhood Chronic Myelogenous Leukemia; Childhood Diffuse Large Cell Lymphoma; Childhood Immunoblastic Large Cell Lymphoma; Childhood Myelodysplastic Syndromes; Childhood Nasal Type Extranodal NK/T-cell Lymphoma; Chronic Myelomonocytic Leukemia; Chronic Phase Chronic Myelogenous Leukemia; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Juvenile Myelomonocytic Leukemia; Mast Cell Leukemia; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Childhood Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Myeloid Leukemia; Recurrent Childhood Anaplastic Large Cell Lymphoma; Recurrent Childhood Grade III Lymphomatoid Granulomatosis; Recurrent Childhood Large Cell Lymphoma; Recurrent Childhood Lymphoblastic Lymphoma; Recurrent Childhood Small Noncleaved Cell Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Recurrent/Refractory Childhood Hodgkin Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Myelodysplastic Syndromes; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Intraocular Lymphoma; Leukemia, Myelomonocytic, Juvenile; Leukemia, Mast-Cell; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence; Leukemia, Hairy Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Alemtuzumab; Whole-Body Irradiation; fludarabine phosphate; Cyclosporine; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (chemotherapy, TBI, transplant) (Experimental): NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive alemtuzumab IV over 6 hours once daily on days -6, -5, and -4 OR days -5 and -4 and fludarabine phosphate IV over 30 minutes on days -4, -3, and -2. Patients also undergo low-dose TBI on day 0.
  ALLOGENEIC PBSCT: After completion of TBI, patients undergo allogeneic PBSCT on day 0.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO or IV every 12 hours on days -3 to 180 followed by a taper until day 365 in the absence of GVHD. Beginning 4-6 hours after completion of allogeneic PBSCT, patients receive mycophenolate mofetil PO every 8 hours on days 0 to 100 followed by a taper until day 156 in the absence of GVHD.
  Interventions: Biological: alemtuzumab; Radiation: total-body irradiation; Drug: fludarabine phosphate; Drug: cyclosporine; Drug: mycophenolate mofetil; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Biological: graft versus host disease prophylaxis/therapy; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: alemtuzumab — Given IV
  Other Names: anti-CD52 monoclonal antibody; Campath-1H; MoAb CD52; Monoclonal Antibody Campath-1H; Monoclonal Antibody CD52
Radiation: total-body irradiation — Undergo low-dose TBI
  Other Names: TBI
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cyclosporine — Given PO or IV
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic stem cell transplantation
Procedure: peripheral blood stem cell transplantation — Undergo PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Biological: graft versus host disease prophylaxis/therapy — Undergo GVHD prophylaxis/therapy
  Other Names: prophylaxis/therapy, graft versus host disease; prophylaxis/therapy, GVHD
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying the side effects and best dose of alemtuzumab when given together with fludarabine phosphate and total-body irradiation followed by cyclosporine and mycophenolate mofetil in treating patients who are undergoing a donor stem cell transplant for hematologic cancer. Giving low doses of chemotherapy, such as fludarabine phosphate, a monoclonal antibody, such as alemtuzumab, and radiation therapy before a donor stem cell transplant helps stop the growth of cancer cells. Giving chemotherapy or radiation therapy before or after transplant also stops the patient's immune system from rejecting the donor's bone marrow stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine which dose of Campath (alemtuzumab) allows related and unrelated human leukocyte antigen (HLA) class-II mismatched hematopoietic cell transplantation (HCT) with an incidence of grade III-IV acute graft-versus-host disease (GVHD) less than 40%.

SECONDARY OBJECTIVES:

I. Incidence of graft rejection.

II. Number of days of steroids >= 1mg/kg required before day 100 in each patient.

III. Incidence of non-relapse mortality.

IV. Risk/incidence of infections.

V. Immune reconstitution.

VI. Risk for disease progression and relapse.

OUTLINE: This is a dose-escalation study of alemtuzumab.

NONMYELOABLATIVE CONDITIONING REGIMEN: Patients receive alemtuzumab intravenously (IV) over 6 hours once daily on days -6, -5, and -4 OR days -5 and -4 and fludarabine phosphate IV over 30 minutes on days -4, -3, and -2. Patients also undergo low-dose total-body irradiation (TBI) on day 0.

ALLOGENEIC PERIPHERAL BLOOD STEM CELL TRANSPLANTATION (PBSCT): After completion of TBI, patients undergo allogeneic PBSCT on day 0.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) or IV every 12 hours on days -3 to 180 followed by a taper until day 365 in the absence of GVHD. Beginning 4-6 hours after completion of allogeneic PBSCT, patients receive mycophenolate mofetil PO every 8 hours on days 0 to 100 followed by a taper until day 156 in the absence of GVHD.

After completion of study treatment, patients are followed up periodically for 12 months, at 18 months, and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be not eligible for conventional transplants and must have disease expected to be stable for at least 100 days without chemotherapy
* Patients with hematologic malignancies treatable with HCT will be included:

  * Aggressive non-Hodgkin lymphomas (NHLs) and other histologies such as diffuse large B-cell NHL: not eligible for autologous HCT, not eligible for conventional myeloablative HCT, or after failed autologous HCT;
  * Low grade NHL: with < 6 month duration of complete response (CR) between courses of conventional therapy;
  * Mantle cell NHL: may be treated in first CR;
  * Chronic lymphocytic leukemia (CLL): must have failed 2 lines of conventional therapy and must be refractory to fludarabine; this includes patients who fail to have a complete or partial response after therapy with a regimen containing fludarabine (or another nucleoside analog] or experience disease relapse within 12 months after completing therapy with a regimen containing fludarabine [or another nucleoside analog);
  * Hodgkin's disease (HD): must have received and failed frontline therapy and have failed or were not eligible for autologous transplant;
  * Multiple myeloma (MM): must have received prior chemotherapy or failed autografting; following a planned autologous transplant [tandem] is allowed;
  * Acute myeloid leukemia (AML): must have < 5% marrow blasts at the time of transplant;
  * Acute lymphocytic leukemia (ALL): must have < 5% marrow blasts at the time of transplant;
  * Chronic myelogenous leukemia (CML): patients will be accepted beyond first clinical progression (CP1) if they have received previous myelosuppressive chemotherapy or HCT, and have < 5% marrow blasts at time of transplant;
  * Myelodysplastic syndrome/myeloproliferative disease (MDS/MPD): must have failed previous myelosuppressive chemotherapy or HCT, and have < 5% marrow blasts at time of transplant;
  * Waldenstrom's macroglobulinemia: must have failed 2 courses of therapy
* Patient refuses to be treated on a conventional transplant protocol; for this inclusion criteria, transplants must be approved by both the participating institution's patient review committee, such as the Patient Care Conference (PCC) at the Fred Hutchinson Cancer Research Center (FHCRC), and the FHCRC principal investigator
* Patient with related or unrelated donors for whom:

  * There is a likelihood of disease progression while HLA typing and results of a preliminary search and the donor pool suggest that a 10/10 HLA-A, B, C, DRB1 and DQB1 matched unrelated donor will not be found;
  * Patient and donor must be matched for at least one DRB1 allele and one DQB1 allele;
  * Best available matches are HLA class I HLA-A, -B, -C allele matched donors allowing for any one or two DRB1 and/or DQB1 antigen/allele mismatch;
  * There is no indication for an autologous transplantation as a treatment option
* DONOR: For HLA matching inclusion criteria, see patient inclusion criteria
* DONOR: Only peripheral blood stem cells (PBSC) will be permitted as a HSC source on this protocol

Exclusion Criteria:

* Positive crossmatch between donor and recipients
* Patient's life expectancy is severely limited by diseases other than malignancy
* Patient has central nervous system (CNS) involvement with disease refractory to intrathecal chemotherapy
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology for patients with AML, ALL or CML
* Patient is a fertile man or woman unwilling to use contraceptives during and for up to 12 months post treatment
* Patient is a female who is pregnant or breastfeeding
* Patient is human immunodeficiency virus (HIV) positive
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers)
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence
* Patient has a fungal infection with radiological progression after receipt of amphotericin B or active triazole for greater than 1 month
* Patient has the following organ dysfunction:

  * Symptomatic coronary artery disease or ejection fraction < 35% or other cardiac failure requiring therapy; ejection fraction is required if age > 50 years or if the patient has a history of anthracyclines or history of cardiac disease;
  * Diffusion capacity of the lung for carbon monoxide (DLCO) < 35% total lung capacity (TLC) < 35%, forced expiratory volume of the lung in one second (FEV1) < 35% and/or receiving supplementary continuous oxygen; the FHCRC study principal investigator (PI) must approve enrollment of all patients with pulmonary nodules;
  * Liver function abnormalities: patient with clinical or laboratory evidence of liver disease will be evaluated for the cause of liver disease, its clinical severity in terms of liver function, bridging fibrosis, and the degree of portal hypertension; the patient will be excluded if he/she is found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3mg/dL, or symptomatic biliary disease
* Patient has poorly controlled hypertension and on multiple antihypertensives
* Karnofsky performance score < 70 for adult patients
* Lansky play-performance score < 70 for pediatric patients
* Patient received cytotoxic agents for "cytoreduction" within three weeks (or the interval in which a cycle of standard chemotherapy would be administered in a non-transplant setting) prior to initiating the nonmyeloablative transplant conditioning; (exceptions are hydroxyurea and imatinib mesylate)
* DONOR: Marrow donors
* DONOR: Positive crossmatch between donor and recipient
* DONOR: Donor is HIV-positive and/or has a medical condition that would result in increased risk for filgrastim (G-CSF) mobilization and harvest of PBSC
* DONOR: Donor age < 12 years

Max Age: 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-03; Primary Completion 2010-07 (Actual); Study Completion 2015-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Sandmaier, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (2):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States
- University of Torino, Torino, Italy

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1 (No Campath): Patients receive fludarabine phosphate IV over 30 minutes on days -4, -3, and -2. Patients also undergo low-dose TBI on day 0.
  Total-body irradiation: Undergo low-dose total-body irradiation
  Fludarabine phosphate: Given IV
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic stem cell transplantation
  Peripheral blood stem cell transplantation: Undergo peripheral blood stem cell transplantation
- Dose Level 2 (40mg Total Dose Campath): Patients receive alemtuzumab IV over 6 hours once daily on days -5 and -4 and fludarabine phosphate IV over 30 minutes on days -4, -3, and -2. Patients also undergo low-dose TBI on day 0.
  Alemtuzumab: Given IV
  Total-body irradiation: Undergo low-dose total-body irradiation
  Fludarabine phosphate: Given IV
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic stem cell transplantation
  Peripheral blood stem cell transplantation: Undergo peripheral blood stem cell transplantation
  NOTE: No subjects were enrolled at this dose level as the escalation rule was not met.
- Dose Level 3 (60mg Total Dose Campath): Patients receive alemtuzumab IV over 6 hours once daily on days -6, -5, and -4 and fludarabine phosphate IV over 30 minutes on days -4, -3, and -2. Patients also undergo low-dose TBI on day 0.
  Alemtuzumab: Given IV
  Total-body irradiation: Undergo low-dose total-body irradiation
  Fludarabine phosphate: Given IV
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic stem cell transplantation
  Peripheral blood stem cell transplantation: Undergo peripheral blood stem cell transplantation
  NOTE: No subjects were enrolled at this dose level as the escalation rule was not met.
Period: Overall Study
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Started | 12 | 0 | 0
Completed | 12 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 2 (40mg Total Dose Campath): Patients receive alemtuzumab IV over 6 hours once daily on days -5 and -4 and fludarabine phosphate IV over 30 minutes on days -4, -3, and -2. Patients also undergo low-dose TBI on day 0.
  Alemtuzumab: Given IV
  Total-body irradiation: Undergo low-dose total-body irradiation
  Fludarabine phosphate: Given IV
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic stem cell transplantation
  Peripheral blood stem cell transplantation: Undergo peripheral blood stem cell transplantation
- Dose Level 3 (60mg Total Dose Campath): Patients receive alemtuzumab IV over 6 hours once daily on days -6, -5, and -4 and fludarabine phosphate IV over 30 minutes on days -4, -3, and -2. Patients also undergo low-dose TBI on day 0.
  Alemtuzumab: Given IV
  Total-body irradiation: Undergo low-dose total-body irradiation
  Fludarabine phosphate: Given IV
  Allogeneic hematopoietic stem cell transplantation: Undergo allogeneic stem cell transplantation
  Peripheral blood stem cell transplantation: Undergo peripheral blood stem cell transplantation
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath) | Total
Number analyzed (Participants) | 12 | 0 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 0 | 0 | 10
  >=65 years | 2 | 0 | 0 | 2
Age, Continuous [Median (Full Range); unit: years] | 58.6 [44 to 71] |  |  | 58.6 [44 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 |  |  | 6
  Male | 6 |  |  | 6
Region of Enrollment [Number; unit: participants]
  United States | 12 |  |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Grade III-IV Acute GVHD
Description: Severity of Individual Organ Involvement
  Liver:
  Stage 2 - bilirubin (3-5.9mg/100ml) Stage 3 - bilirubin (6-14.9mg/100ml) Stage 4 - bilirubin > 15mg/100ml
  Gut:
  Diarrhea is graded stage 1 to stage 4 in severity. Nausea and vomiting and/or anorexia caused by GVHD is assigned as stage 1 in severity. The severity of gut involvement is assigned to the most severe involvement noted. Patients with visible bloody diarrhea are at least stage 2 gut and grade 3 overall
  Severity of GVHD
  Grade III - Stage 2 to 4 gastrointestinal involvement and/or Stage 2 to 4 liver involvement with or without a rash Grade IV - Pattern and severity of GVHD similar to grade 3 with extreme constitutional symptoms or death
Time Frame: 100 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Number analyzed (Participants) | 12 | 0 | 0
percentage of participants | 25 |  |

2. Secondary Outcome: Incidence of Graft Rejection
Description: Percentage patients that experienced graft rejection.
Time Frame: 84 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Number analyzed (Participants) | 12 | 0 | 0
percentage of participants | 0 |  |

3. Secondary Outcome: Incidence of High-dose Corticosteroid Utilization.
Description: Percentage patients requiring steroids greater than 1 mg/kg.
Time Frame: 100 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Number analyzed (Participants) | 12 | 0 | 0
percentage of participants | 83.3 |  |

4. Secondary Outcome: Incidence of Non-relapse Mortality
Description: Percentage patient deaths due to non-relapse mortality
Time Frame: 100 days after transplant
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Number analyzed (Participants) | 12 | 0 | 0
percentage of participants | 8.3 |  |

5. Secondary Outcome: Incidence of Infection
Description: Percentage patients that experienced infection(s).
Time Frame: Up to 5 years post-transplant
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Number analyzed (Participants) | 12 | 0 | 0
percentage of participants | 100 |  |

6. Secondary Outcome: Immune Reconstitution
Description: The outcome of immune reconstitution was not analyzed by the collaborating laboratory because only a small number of patients were only enrolled in Dose Level 1 (no alemtuzumab). The Dose Level 1 patients were going to be the baseline for which to compare the other patients on Dose Level 2 (and 3) who would have received alemtuzumab. The collaborating investigator determined that the study was not worthwhile performing based on this information.
Time Frame: Up to 1 year post-transplant
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Disease Progression/Relapse
Description: CML New cytogenetic abnormality and/or development of accelerated phase or blast crisis. The criteria for accelerated phase will be defined as unexplained fever greater than 38.3°C, new clonal cytogenetic abnormalities in addition to a single Ph-positive chromosome, marrow blasts and promyelocytes >20%.
  AML, ALL >5% marrow blasts by morphologic or flow cytometric, or appearance of extramedullary disease.
  CLL ≥1 of: Physical exam/Imaging studies (nodes, liver, and/or spleen) ≥50% increase or new, circulating lymphocytes by morphology and/or flow cytometry ≥50% increase, and lymph node biopsy w/ Richter's transformation.
  NHL >25% increase in the sum of the products of the perpendicular diameters of marker lesions, or the appearance of new lesions.
  MM
  ≥100% increase of the serum myeloma protein from its lowest level, or reappearance of myeloma peaks that had disappeared w/ treatment; or definite increase in the size or number of plasmacytomas or lytic bone lesions.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Number analyzed (Participants) | 12 | 0 | 0
percentage of participants | 25 |  |

ADVERSE EVENTS:
Time Frame: AEs: Conditioning through Day 100; SAEs: Conditioning through Day 200
Arm/Group | Dose Level 1 (No Campath) | Dose Level 2 (40mg Total Dose Campath) | Dose Level 3 (60mg Total Dose Campath)
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 7/12 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (No Campath) (N=12) | Dose Level 2 (40mg Total Dose Campath) (N=0) | Dose Level 3 (60mg Total Dose Campath) (N=0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Concurrent elevated bilirubin. Patient expired
Death due to GVHD (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1 (No Campath) (N=12) | Dose Level 2 (40mg Total Dose Campath) (N=0) | Dose Level 3 (60mg Total Dose Campath) (N=0)
Acute coronary syndrome (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 4 (4) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes